CLINICAL TRIAL: NCT00755742
Title: Evaluation of the Impact of a Combined Program of Diet, Exercise and Behavior Modification on the Insulin Resistance and Adipokine Profile in Obese Patients With Current and Cured Chronic Hepatitis C.
Brief Title: Lifestyle Intervention Targetting Obesity and Insulin Resistance in Chronic Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Venessa Pattullo, Research Collaborator, University Health Network, Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0545-AE
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Obesity; Insulin Resistance; Metabolic Syndrome; Hepatitis C
Keywords: obesity; insulin resistance; metabolic syndrome; hepatitis C; adipokine; TNF; leptin; adiponectin; fatigue; mood; depression; exercise; diet; counseling; behavior modification
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome; Hepatitis C; Fatigue; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - Viremic / Non-cirrhotic (Experimental): 13 obese and insulin resistant, non-cirrhotic, non-diabetic (by fasting glucose), non-genotype 3 patients with chronic hepatitis C (HCV RNA positive) will undergo 24 week lifestyle intervention comprising diet, physical activity (monitored by pedometers) in combination with behavior modification counseling. This arm includes patients who are naive to antiviral therapy, relapsed or not responded to antiviral therapy.
  Interventions: Other: Lifestyle intervention
- Group 2 - Non-viremic / Non-cirrhotic (Active Comparator): 13 obese and insulin resistant, non-cirrhotic, non-diabetic (by fasting glucose), non-genotype 3 patients with cured chronic hepatitis C (HCV RNA negative) will undergo 24 week lifestyle intervention comprising diet, physical activity (monitored by pedometers) in combination with behavior modification counseling. This arm includes patients who have cleared hepatitis C virus with previous antiviral therapy.
  Interventions: Other: Lifestyle intervention
- Group 3 - Viremic / Cirrhotic (Experimental): 13 obese and insulin resistant, cirrhotic, non-diabetic (by fasting glucose), non-genotype 3 patients with chronic hepatitis C (HCV RNA positive) will undergo 24 week lifestyle intervention comprising diet, physical activity (monitored by pedometers) in combination with behavior modification counseling. This arm includes patients who are naive to antiviral therapy, relapsed or not responded to antiviral therapy.
  Interventions: Other: Lifestyle intervention
- Group 4 - Non-viremic / Cirrhotic (Active Comparator): 13 obese and insulin resistant, cirrhotic, non-diabetic (by fasting glucose), non-genotype 3 patients with cured chronic hepatitis C (HCV RNA negative) will undergo 24 week lifestyle intervention comprising diet, physical activity (monitored by pedometers) in combination with behavior modification counseling. This arm includes patients who have cleared hepatitis C virus with previous antiviral therapy
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — The 3-pronged lifestyle intervention is designed to deliver a period of intensive contact (week 0-12) and less-intensive contact (weeks 12-24):
  i) Behavior Modification Counseling: The principles of motivational enhancement and cognitive-behavior therapy (MET/CBT) will be utilized at each visit and telephone contact to provide individually tailored counseling. The goal is to enhance internal motivation and facilitate changes in lifestyle that are adaptable to each participant's usual habits.
  ii) Physical activity target: increment in activity of at least 3000 steps/day above the baseline, or total activity of 10,000 steps/day (whichever is greater).
  iii) Dietary assessment and nutritional plan: A diet plan designed to both lose weight and improve insulin resistance will be provided.

SUMMARY:
Chronic hepatitis C (CHC) infection affects approximately 1 in 100 Canadians. Untreated, CHC has significant long-term consequences including cirrhosis, liver cancer and liver failure. CHC is intrinsically linked to both obesity and insulin resistance (IR) or "pre-diabetes", their co-existence worsens overall health outcomes. We have demonstrated that obesity (BMI ≥30kg/m2) is over twice as common amongst patients with CHC (28.8%) compared with the general Canadian population. Obesity superimposed on CHC reduces the success of antiviral treatment and promotes liver scarring (hepatic fibrosis), fatty liver (steatosis) and increases the risk of liver cancer. Both CHC and obesity contribute to IR putting these patients at risk of type 2 diabetes. IR, like obesity in CHC, reduces antiviral success rates. We have shown that diabetics are at higher risk of developing liver cancer compared with non-diabetics. It is therefore timely to address lifestyle modification to delay the onset of diabetes. We will examine the impact of a multidisciplinary lifestyle program on the insulin resistance in 52 obese "pre-diabetic" patients with current or past CHC. The 24 week program comprises an individualized nutritional and exercise plan supported by behavior modification counseling. Through gaining a better understanding of links between obesity, insulin resistance and hepatitis C infection we hope to delay the onset of diabetes and reduce the likelihood of all their untoward effects on the liver.

DETAILED DESCRIPTION:
The hepatitis C virus (HCV) chronically infects an estimated 240,000 in Canada and 170 million worldwide. Untreated, CHC is associated with significant long-term clinical consequences including cirrhosis, liver failure and hepatocellular cancer (HCC), and it is the most common indication for liver transplantation in North America. CHC is associated with metabolic manifestations independent of the degree of hepatic fibrosis which include insulin resistance (IR) and type 2 diabetes (T2DM), which have a significantly higher prevalence in CHC compared with the general population. Patients with CHC and T2DM have an increased risk of HCC in addition to morbidity from systemic complications.

Our previous work demonstrates that the prevalence of obesity (BMI ≥30kg/m2) amongst patients with CHC is 28.8%, over twice the prevalence in the Canadian population, and the presence of obesity is independently associated with viremia (positive HCV-RNA). Obesity promotes hepatic fibrosis progression and is independently associated with IR in non-cirrhotic CHC; the prevalence of IR increases with higher BMI in CHC. Insulin resistance can be reversed if viral clearance is achieved; however loss of IR is less likely to occur in the obese even if they have cleared the virus. Obesity and IR are associated with non-response to antiviral therapy. Whilst IR has been improved with the use of metformin in patients with CHC, this was ineffective in increasing rates of response to antiviral treatment. The aims of our study are:

1. To evaluate the effect of a three-pronged lifestyle intervention comprising diet, exercise and behavior modification on insulin resistance in obese patients with current and cured chronic hepatitis C.
2. To formulate specific recommendations for lifestyle changes to improve insulin resistance and lose weight, thereby reducing the risk of diabetes and other metabolic complications, and potentially enhancing response to antiviral therapy in obese patients with CHC.
3. To examine the impact of this intervention on IR, insulin sensitivity and serum adipokine levels for the purpose of investigating the mechanism of insulin resistance in obesity with and without viremia due to chronic hepatitis C infection.

We will utilize a multidisciplinary approach by collaborating with the disciplines of gastroenterology, nutrition, endocrinology, exercise physiology and psychiatry. This prospective study will include 13 non-cirrhotic and 13 cirrhotic, insulin resistant (HOMA-IR ≥2.1) and obese patients (non-Genotype 3, as the latter have marked fatty liver in absence of obesity); as well as 13 non-cirrhotic and 13 cirrhotic, insulin resistant and obese patients with successfully treated CHC (ie now non-viremic) to act as controls. Assessments for measures of IR and obesity (including oral glucose tolerance test to calculate insulin sensitivity index (ISI), serum adipokines, free fatty acids, anthropometry and body composition by abdominal DEXA) will be made. The HOMA-IR (measuring hepatic IR) will be the primary outcome for the experimental maneuver, which will take place over 24 weeks. It will comprise 3 components:

1. Diet: participants will be advised on an individually tailored diet of low glycemic foods, low total fat (but rich in omega-3 fatty acid) and high fiber aimed at both weight loss and improvement of insulin resistance.
2. Exercise: physical activity will be measured with the use of a personal pedometer, and participants given a step target of 10000 steps per day, or an increment of 3000 steps per day from their baseline activity (whichever is greater).
3. Behavior Modification: the change in diet and physical activity will be facilitated by a 12-week face-to face program followed by a 12-week telephone program based on the principals of motivational interviewing and behavior theory.

The intercurrence of obesity and IR in subjects chronically infected with hepatitis C exacerbates their poor current and future health status. As the pathophysiology of IR in patients with CHC may differ from those who are obese but no longer infected, we will quantify the benefits of the lifestyle intervention in these two patient groups as gauged by fall in HOMA-IR score and improvement in ISI. Our long-term goals are to improve the outcome of antiviral therapy and reduce the burden of CHC, obesity and type 2 diabetes related morbidity. This we hope to achieve through gaining a better understanding of the mechanisms involved in the development of IR in the obese with and without current CHC.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI >/= 30)
* insulin resistant (HOMA-IR >/= 2.1)

Exclusion Criteria:

* Genotype 3 patients
* Women with ongoing pregnancy or who are breast-feeding
* Patients with any other other underlying liver disease (viral, alcoholic, druginduced, autoimmune, metabolic, genetic).
* Patients currently on antiviral therapy, or who have ceased therapy within 6 months of recruitment to the study.
* Patients with other causes for insulin resistance e.g., excess counter-regulatory hormones: glucocorticoids, catecholamines, growth hormone, polycystic ovary syndrome).
* Patients on steroids or other drug that affects insulin resistance, which are unable to be stopped for 3 days prior to IR testing.
* Patients with overt diabetes (based on results of fasting plasma glucose) will be excluded from participation as we are focusing on insulin resistance in the absence of diabetes.
* Conditions which preclude a sudden increase in physical activity:

  * History or other evidence of chronic pulmonary disease associated with functional limitation.
  * History of severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases).
  * Unable to 10000 steps/day eg physical disability, morbid obesity.
* Evidence of ongoing substance use (including alcohol consumption >20g/day for men and >10g/day for women) within one year of study recruitment.
* Poor veins (inadequate venous access)
* Inability or unwillingness to provide informed consent or abide by study requirements eg severe psychiatric illness, lives remotely, time commitment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 12 and 24 weeks

SECONDARY OUTCOMES:
TNF-alpha | 12 and 24 weeks
leptin | 12 and 24 weeks
adiponectin | 12 and 24 weeks
fatigue score | 12 and 24 weeks
mood score | 12 and 24 weeks
cholesterol | 12 and 24 weeks
triglycerides | 12 and 24 weeks
HDL-cholesterol | 12 and 24 weeks
LDL-cholesterol | 12 and 24 weeks
RBC fatty acid composition | 12 and 24 weeks
BMI | 12 and 24 weeks
Waist circumference | 12 and 24 weeks
Metabolic Syndrome | 12 and 24 weeks
CLDQ (Chronic Liver Disease Questionnaire) | 12 and 24 weeks
Liver and Peripheral Insulin Resistance | 12 and 24 weeks
  Scores derived from glucose and insulin levels in the oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Heathcote, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada